CLINICAL TRIAL: NCT06895317
Title: Chronic Low Back Pain: Innovative E-healTh DiagnOstics and RehabiliTation Towards an IntegrAted and PersonaLized SPINE Care (TOTALSPINE) - UO04
Brief Title: Chronic Low Back Pain: TOTALSPINE - UO04
Acronym: TOTALSPINE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Collaborators: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Francesco Corallo, Executive Psychologist, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 181.24 CET2 cbm; PNRR-MCNT2-2023-12378359 (Other Grant/Funding Number: ITALIAN MINISTRY OF HEALTH)
Record Dates: First submitted 2025-02-27; First posted 2025-03-26 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-08

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: Chronic low back pain; quality of life; chronic pain; treatment adherence; anxiety; depression; neuropsychological; psychosocial assessment
MeSH Terms: conditions — Chronic Pain; Treatment Adherence and Compliance; Anxiety Disorders; Depression | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote rehabilitation (Experimental): Remote therapy will be delivered for the experimental group to test the effectiveness of remote physiotherapy rehabilitation
  Interventions: Behavioral: Remote rehabilitation
- Face-to-face rehabilitation (Active Comparator): For the control group, traditional face-to-face therapy will be delivered to test the difference with remote physiotherapy rehabilitation
  Interventions: Behavioral: Rehabilitation face to face

INTERVENTIONS:
Behavioral: Remote rehabilitation — To develop and validate a quantitative assessment system based on wearable sensors
  Other Names: Face to face rehabilitation
  Arms: Remote rehabilitation
Behavioral: Rehabilitation face to face — Compare the validity of face-to-face physiotherapy with remote physiotherapy
  Arms: Face-to-face rehabilitation

SUMMARY:
Background: Low back pain (LBP) is the primary factor contributing to years lived with disability. In view of the close correlation between the functions of the body, which cannot be examined piecemeal but as an integrated system, a holistic approach allows for a comprehensive assessment of the patient. The goal of our protocol is to identify all psychosocial risk factors that could worsen the patient's condition at the time of diagnosis by examining all possible related dimensions: cognitive function, anxiety and depression, pain perception, treatment adherence, the sexual sphere, family dynamics, social support, dysfunctional communication, quality of life while also considering attribution of causes.

Methods: At least 86 patients will participate in the survey. At T0, they will undergo neuropsychological, psychological and associated clinical condition assessment through standardized tests and ad hoc questionnaires. After 1 month (T1), 2 months (T2) and 6 months (T3), the same tests will be repeated.

Expected results: We expect this study to provide a comprehensive, in-depth, and integrated understanding of the patient, shedding light on the challenges they may face in managing chronic low back pain.

Repeated administration of the questionnaires will allow us to monitor the patient over time, assess any changes in their health status, and structure an intervention tailored to their needs.

Conclusions: By emphasizing these often neglected areas through a comprehensive, multi-step assessment, it will be possible to quantify and analyze how these risk factors can affect patients' well-being and hinder the treatment process and recovery.

DETAILED DESCRIPTION:
1. Introduction Low back pain (LBP) is the primary factor contributing to years lived with disability.

Non-specific LBP is defined as LBP not attributable to a known cause and accounts for 90-95% of LBP cases.

The estimated prevalence of non-specific LBP is 18%. The prognosis for LBP is not as good as previously thought, particularly due to the frequent relapses or the transition to chronic LBP. One of the reasons is the hardworkingness of the mechanisms involved in chronic back pain. Despite the high prevalence of back pain and the enormous personal and social costs, the response of the healthcare system has not been satisfactory. The traditional biomedical approach to back pain has been particularly inadequate. Since social and psychological factors are involved in the pathogenesis of chronic back pain, assessing the patient's condition is not a simple task. This condition, in fact, significantly affects individuals' daily lives.

Therefore, effective strategies play an important role in minimizing the impact of LBP.

The failure of the biomedical model to produce better outcomes for chronic back pain has led to the adoption of a biopsychosocial model. The existence of psychosocial factors negatively impacts the outcomes of LBP and contributes to its chronicity. The biopsychosocial model provides a framework to explain the complexity of disabling LBP through a multidimensional clinical approach, incorporating the interaction between the social, psychological, and biological dimensions of pain, context, and behavioral conditioning.

A predominantly quantitative line of research shows that individuals suffering from chronic pain are subject to job loss, socioeconomic deprivation, subsequent depression, and social isolation. Patients with chronic pain have higher rates of depression compared to the general population, and many of those with chronic LBP (CLBP) endure distressing experiences characterized by catastrophization, passive coping, low self-efficacy, and high levels of anxiety, which are thought to predict and maintain chronicity.

Psychological risk factors for an unfavorable prognosis can be clinically identified and addressed within interventions. Kendall et al., 1998 coined the term "yellow flags" to understand the psychological risk factors and social and environmental risk factors for prolonged disability and failure to return to work as a consequence of musculoskeletal symptoms caused by LBP. These psychological risk factors included fears of pain or injury, unhelpful beliefs about recovery, and distressed affect (e.g., despair and anxiety).

Social and environmental risk factors included workers' perceptions that the workplace is unsupportive and that the care provided is unsatisfactory.

More recently, a distinction has been made between psychological risk factors that could be considered "normal" but unhelpful psychological reactions to musculoskeletal symptoms (e.g., the belief that pain necessarily implies damage) and "abnormal" psychological or psychiatric factors or disorders (e.g., post-traumatic stress disorder, major depression) that suggest a diagnosable psychopathology. The psychological reactions defined as "normal" should be described as yellow flags, while those that meet the criteria for psychopathology should be termed orange flags.

The primary significance of this distinction is to differentiate yellow flag factors, which may be amenable to short-term psychological intervention, from orange flag factors that require long-term psychological intervention.

Early identification of these factors may be key to structuring more effective interventions to reduce or prevent chronic or recurring disability. Moreover, since LBP imposes a significant economic burden on healthcare systems, it may be more cost-effective to address a broader target population early with simple, low-cost interventions rather than spending extensive time and resources rehabilitating a smaller group of patients with back pain who have become disabled due to chronic pain.

Early active management of LBP is indeed a useful strategy to reduce the risk of transition to CLBP.

Leveraging digital platforms, wearable sensors, and artificial intelligence, an innovative solution emerges to enable a personalized and integrated approach to the diagnosis and rehabilitation of CLBP.

These technologies have the potential to revolutionize care delivery, providing personalized interventions and improving patient outcomes. The latest technological innovations in fact can contribute to early screening and especially to intervention delivered even at a distance that is usable to a large part of the population, making not only diagnosis but treatment more accessible, promoting a positive prognosis and more functional pain management, so that a good quality of life is safeguarded and preserved. As a multifactorial pathogenesis underlying the disorder is recognized, it is also important to educate the patient to modify the negative aspects that negatively affect their condition. Modifiable, lifestyle-related risk factors include, first and foremost, cigarette smoking and obesity. Both are associated with both the development and persistence of the disorder. Professional risk factors, such as lifting heavy loads, prolonged maintenance of incorrect postures, and continuous exposure to vibrations, also seem to play a significant role.

Not only physical stress in the strict sense, but also emotional stress that can arise from job dissatisfaction or economic and/or social factors can contribute to the development and persistence of LBP.

It is important to establish an effective therapeutic relationship right from the start, which helps the patient understand that they are embarking on a different path where they must also be an active participant in their care. Indeed, the patient, with the help and support of professionals, can mobilize latent strengths and resources to establish an alliance and pursue a shared goal.

This article describes the research project "Chronic low back pain: Innovative e-healTh diagnOstics and rehabiliTation toward integrAted and personaLized SPINE (TOTALSPINE) care (PNRR-MCNT2-2023-12378359)." This paper outlines the design and methodology of the component related to our operational unit focused on neuropsychological assessment. Given the strong correlation between the development and outcomes of the disease and the numerous interconnected factors, which cannot be assessed in isolation but rather as part of an integrated system, the overarching goal of this research project is to develop and validate innovative tools for comprehensive, yet personalized clinical assessment. Ultimately, these tools aim to facilitate the delivery of effective treatments for patients with chronic low back pain (CLBP).

Part of the research project is devoted to understanding whether an e-Health-based rehabilitation protocol delivered through a mobile application can improve disability and other health-related outcomes like traditional face-to-face rehabilitation treatment in an RCT on patients with CLBP.

This purpose is related to our role as an operating unit, whose task is to evaluate the patient before and after treatment to examine the effects and possible validation and promotion of rehabilitation treatment delivered remotely. In particular, this article focuses on the part of the project related to the evaluation of the patient's overall functioning. The psychosocial assessment will indeed include all areas affected by the condition of chronic pain, all contexts in which the patient is involved, and all aspects that are negatively and persistently impacted by the pathology, contributing to a reduced quality of life.

This is to gain a holistic view of the patient's health.

The specific objectives of our operational unit in the project are as follows:

1. Evaluation of the psychological aspects of LBP before and after treatment
2. Assessment of functional status
3. Evaluation of cognitive performance
4. Assessment of mood and related psychopathologies
5. Evaluation of health-related quality of life
6. Assessment of social support
7. Evaluation of sleep quality
8. Assessment of the burden of comorbidity
9. Evaluation of treatment adherence

These dimensions will be assessed through a specific battery of tests:

* Pain Self Efficacy Questionnaire (PSEQ)
* Oswestry Disability Index (ODI)
* Pain Catastrophizing Scale (PCS)
* 12-Item Short Form Survey (SF-12) or 36-Item Short Form Survey (SF-36)
* Beck's Anxiety Inventory (BAI)
* Center for Epidemiologic Studies - Depression Scale (CES-D)
* Patient Health Engagement Scale (PHE-s)
* The Montreal Cognitive Assessment (MoCA)
* Two specially designed questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* CLBP of discogenic origin rated above 4 on the Numeric Rating Scale (NRS) in the 2 weeks prior, ongoing for the last 6 weeks up to 12 months before inclusion

Exclusion Criteria:

* Past or present medical history of "red flags" (e.g., cancer, fractures, infections) or specific causes of non-discogenic LBP; 2) Having received physical therapy for LBP in the last 6 months;
* Previous spinal surgery;
* Severe or progressive neurological deficits;
* Any serious medical comorbidity that, in the opinion of the Principal Investigator (PI), would make participation unsafe or impossible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
psychosocial assessment through the use of tests to assess the extent of pain | At the enrollment stage before the start of treatment
  The Pain Self-Efficacy Questionnaire (PSEQ), will be used to assess how patients maintain their autonomy despite perceived pain. This among the various measures that will be used is considered primary outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Irccs Centro Neurolesi Bonino Pulejo, Messina, Italy
  - Campus Biomedico Roma, Roma, IT

IPD SHARING:
Plan to Share IPD: No
The personal data (IPD) that will be collected in this study are not available openly for sensitivity reasons and are available from the clinical trial protocol scientific officer upon reasonable request.

REFERENCES:
- [Derived] Anselmo A, Pagano M, Corallo F, Cappadona I, Cardile D, Russo F, Laudisio A, Papalia GF, Quartarone A, Calabro RS. Psychosocial Assessment as a Key Component in an Integrated, Personalized Care Pathway: A Protocol for a Low Back Pain Randomized Controlled Trial. Pain Ther. 2025 Jun;14(3):1155-1168. doi: 10.1007/s40122-025-00741-7. Epub 2025 Apr 29. PMID 40299187